CLINICAL TRIAL: NCT00847899
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Exploratory, 28-Day Study to Examine the Effects of AR9281 on Blood Pressure and Glucose Tolerance in Patients With Mild to Moderate Hypertension and Impaired Glucose Tolerance
Brief Title: Evaluation of Soluble Epoxide Hydrolase (s-EH) Inhibitor in Patients With Mild to Moderate Hypertension and Impaired Glucose Tolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arete Therapeutics (Industry)
Responsible Party: Calvert Lee, Sr. CRA, Arete Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AR9281-CLN-003
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Hypertension; Impaired Glucose Tolerance
Keywords: hypertension; impaired glucose tolerance; s-EH enzyme inhibition; pre-diabetes
MeSH Terms: conditions — Hypertension; Glucose Intolerance | interventions — 1-(1-acetyl-piperidine-4-yl)-3-adamantan-1-yl-urea

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): AR9281
  Interventions: Drug: AR9281
- 2 (Active Comparator): AR9281
  Interventions: Drug: AR9281
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AR9281 — AR9281 taken in BID dosing regimen for 28 days
  Arms: 1
Drug: AR9281 — AR9281 taken in TID dosing regimen for 28 days
  Arms: 2
Drug: Placebo — Placebo taken in BID dosing regimen for 28 days
  Arms: 3
Drug: Placebo — Placebo taken in TID dosing regimen for 28 days
  Arms: 4

SUMMARY:
The purpose of this study is to determine the safety and efficacy of AR9281, a novel s-EH enzyme inhibitor, in improving glucose metabolism and blood pressure in patients with impaired glucose tolerance and mild to moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* mild to moderate hypertension
* naive to antihypertensive medication or on two or less antihypertensive medications
* impaired glucose tolerance
* mild obesity

Exclusion Criteria:

* Diagnosis of Type 1 or Type 2 diabetes
* History of severe heart failure
* AST, ALT levels more than twice the normal range

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Systolic and Diastolic blood pressure | 28 day treatment period
Glucose dynamics and insulin sensitivity | 28 day treatment period

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - Arete Investigational site, Mobile, Alabama
  - Arete Investigational site, Muscle Shoals, Alabama
  - Arete Investigational site, Anaheim, California
  - Arete Investigational site, Concord, California
  - Arete Investigational site, Mission Hills, California
  - Arete Investigational site, Bradenton, Florida
  - Arete Investigational site, DeLand, Florida
  - Arete Investigational site, Jacksonville, Florida
  - Arete Investigational site, Largo, Florida
  - Arete Investigational site, Miami, Florida
  - Arete Investigational site, New Port Richey, Florida
  - Arete Investigational site, Pembroke Pines, Florida
  - Arete Investigational site, Port Orange, Florida
  - Arete Investigational site, Tampa, Florida
  - Arete Investigational site, Marietta, Georgia
  - Arete Investigational site, Addison, Illinois
  - Arete Investigational site, Louisville, Kentucky
  - Arete Investigational site, Brockton, Massachusetts
  - Arete Investigational site, Paw Paw, Michigan
  - Arete Investigational site, Las Vegas, Nevada
  - Arete Investigational site, Cincinnati, Ohio
  - Arete Investigational site, Marion, Ohio
  - Arete investigational site, Mount Gilead, Ohio
  - Arete Investigational site, Oklahoma City, Oklahoma
  - Arete Investigational site, Eugene, Oregon
  - Arete Investigational site, Austin, Texas
  - Arete Investigational site, Dallas, Texas
  - Arete Investigational site, San Antonio, Texas
  - Arete Investigational site, Orem, Utah

REFERENCES:
- See also: Arete Therapeutics home website — http://www.aretetherapeutics.com